CLINICAL TRIAL: NCT00350298
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled Study of the Clinical Effectiveness of a Human Monoclonal Antibody to Clostridium Difficile Toxin A (GS-CDA1) and a Human Monoclonal Antibody to Clostridium Difficile Toxin B (MDX-1388) in Patients Being Treated for Clostridium Difficile Associated Disease
Brief Title: Study of the Clinical Effectiveness of a Human Monoclonal Antibody to C. Difficile Toxin A and Toxin B in Patients With Clostridium Difficile Associated Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MassBiologics (Other)
Collaborators: Medarex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA-GCDX-06-02
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Results first posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Clostridium Infections
Keywords: Monoclonal antibody,; Clostridium difficile Associated Diarrhea
MeSH Terms: conditions — Clostridium Infections | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GS-CDA1/MDX-1388 (Experimental): Biological: GS-CDA1/MDX-1388 One Intravenous dose
  Interventions: Biological: GS-CDA1/MDX-1388
- Placebo (Placebo Comparator): Biological: normal saline (0.9% sodium chloride) One Intravenous dose
  Interventions: Biological: normal saline

INTERVENTIONS:
Biological: GS-CDA1/MDX-1388 — One Intravenous dose
  Arms: GS-CDA1/MDX-1388
Biological: normal saline — One Intravenous dose
  Arms: Placebo

SUMMARY:
Patients with Clostridium difficile associated disease who fulfill the eligibility criteria will be approached to participate. All study patients must receive standard of care treatment for Clostridium difficile associated disease. Enrolled patients will be randomized to receive a single intravenous solution of a human monoclonal antibody (huMab) to C. difficile toxin A (GS-CDA1) combined with a human monoclonal antibody to C. difficile toxin B (MDX-1388) or 0.9% sodium chloride as placebo in a 1:1 treatment allocation. Patients will be evaluated for safety and clinical outcomes through day 84 +/- 10 days. Occurrence of adverse events, use of concomitant medications, and stool output will be assessed at scheduled phone contacts and study visits. Some patients enrolled will have a subsequent visit on day 168 ± 14 days.

DETAILED DESCRIPTION:
This study is a phase II, randomized, double-blind, placebo-controlled study in patients diagnosed with Clostridium difficile associated disease. Patients with Clostridium difficile associated disease will be identified either from stool test results or by physician referral, and those who fulfill the eligibility criteria will be approached to participate. All study patients must receive standard of care treatment for Clostridium difficile associated disease. Enrolled patients will be randomized to receive a single intravenous solution of a human monoclonal antibody to C. difficile toxin A (GS-CDA1) combined with a human monoclonal antibody to C. difficile toxin B (MDX-1388) or 0.9% sodium chloride as placebo in a 1:1 treatment allocation. One hundred patients will be enrolled in the combination monoclonal antibody treated arm and 100 patients will be enrolled in the placebo arm. Patients will be evaluated through day 84 ± 10 days after receipt of study infusion for safety and clinical outcomes. Blood samples for safety analyses, anti-toxin A and anti-toxin B antibody measurements and human anti-human antibody (HAHA) titers will be collected at scheduled times. Study visits will occur on days 3 ± 1, 10 ± 2, 28 ± 3, 56 ± 7 and on day 84 ± 10 days. Occurrence of adverse events, use of concomitant medications, and record of stool output will be assessed at scheduled phone contacts and study visits. The first 20 patients enrolled will have a subsequent visit on day 168 ± 14 days for an additional blood collection for HAHA analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient > 18 years of age with diarrhea associated with a positive stool test for C. difficile toxin(s). Patients may be diagnosed with C. difficile by hospital/clinic/reference microbiology laboratory test or by a rapid diagnostic test performed by the study staff and positive test result must be within 14 days of enrollment.
2. Patient must receive standard of care treatment for C. difficile associated disease. Standard of care treatment should include either metronidazole by mouth or intravenously or vancomycin by mouth.
3. Patient or legal representative must have read, understood, and provided written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization after the nature of the study has been fully explained.

Exclusion Criteria:

1. History of chronic diarrheal illness such as ulcerative colitis or Crohn's disease.
2. Score of 4 on modified Horn's index
3. Severe C. difficile colitis with planned surgery in less than 24 hours.
4. Positive pregnancy test within 24 hours of study infusion or an unwillingness to undergo pregnancy testing in females of child-bearing potential. Females capable of child-bearing must agree not to become pregnant from the time of study enrollment until at least 3 months after completion of study infusion. If a woman is sexually active and has no history of hysterectomy or tubal ligation, she must agree to use hormonal or barrier birth control with spermicidal gel.
5. Breastfeeding.
6. Receipt of other investigational study agent within previous 30 days.
7. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of the patient participating in the study or make it unlikely the patient could complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-07-20 (Actual); Primary Completion 2008-06-25 (Actual); Study Completion 2008-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Baxter, MD, Principal Investigator — Kaiser Permanente; Herbert DuPont, MD, Principal Investigator — St. Lukes Episcopal Hospital, Houston, TX; Joseph White, MD, Principal Investigator — Scott and White Memorial Hospital, Temple, TX; David Chen, MD, Principal Investigator — MultiCare Health System Research Services, Tacoma, WA; Jorge Reyno, MD, Principal Investigator — Rapid City Regional Hospital, Rapid City, SD; Henry S. Sacks, MD, PhD, Principal Investigator — Mount Sinai Hospital, New York, NY; Charles N. Bernstein, MD, Principal Investigator — University of Manitoba, Health Sciences Centre, Winnepeg, Manitoba, Canada; Michael J. Tan, MD, Principal Investigator — Summa Health Systems, Akron, Ohio; Michael C. Meadors, MD, Principal Investigator — All-Trials Clinical Research, LLC, Winston-Salem, NC; Ian M. Baird, MD, Principal Investigator — Remington-Davis Clinical Research; Andre Poirier, MD, MSc, Principal Investigator — Centre Hospitalier Regional de Trois-Rivieres; Martha I. Buitrago, MD, Principal Investigator — Idaho Falls Infectious Diseases, PLLC; Thomas Kovacs, MD, Principal Investigator — UCLA CURE Digestive Diseases Research Center; Alfred Bacon, MD, Principal Investigator — Christiana Care Health Systems; Kathleen Casey, MD, Principal Investigator — Jersey Shore University Medical Center; C. Douglas Cochran, MD, Principal Investigator — St. Luke's Hospital, Kansas City, Missouri; Donald Daly, MD, Principal Investigator — Vancouver Island Health Research Centre; Anil Dhar, MBBS, Principal Investigator — Windsor Regional Hospital; Gerald Evans, MD, Principal Investigator — Kingston Health Sciences Centre; Richard Greenberg, MD, Principal Investigator — University of Kentucky; Thomas Louie, MD, Principal Investigator — University of Calgary Foothills Medical Center; Thomas Nowak, MD, Principal Investigator — Central Indiana Gastroenterology Group; Jose Prieto, MD, Principal Investigator — Dr. Kiran C. Patel Research Institute; Daniel Schroeder, MD, Principal Investigator — Chest, Infectious Diseases and Critical Care Assoc., PC; Ann Silverman, MD, Principal Investigator — Henry Ford Health System; John Pullman, MD, Principal Investigator — Mercury Street Medical Group; Rodney J Mason, MD, Principal Investigator — LAC+USC Medical Center; Doria Grimard, MD, Principal Investigator — Centre de Sante et de Services Sociaux de Chicoutimi; Darrell Pardi, MD, Principal Investigator — Mayo Clinic
Locations (29):
- United States (22):
  - LAC/USC Medical Center, Los Angeles, California
  - UCLA CURE Digestive Diseases Center, Los Angeles, California
  - Kaiser Permanente Vaccine Study Center, Oakland, California
  - Christiana Care Health Systems, Newark, Delaware
  - Dr. Kiran C. Patel Research Institute, Tampa, Florida
  - Idaho Falls Infectious Diseases, PLLC, Idaho Falls, Idaho
  - Central Indiana Gastroenterology Group, Anderson, Indiana
  - Chest, Infectious Diseases and Critical Care Assoc., PC, Des Moines, Iowa
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Henry Ford Health System, West Bloomfield, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint James Healthcare, Butte, Montana
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Mount Sinai Hospital, New York, New York
  - All-Trials Clinical Research, LLC, Winston-Salem, North Carolina
  - Summa Health System, Akron, Ohio
  - Remington-Davis Clinical Research, Columbus, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - St. Lukes Episcopal Hospital, Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - MultiCare Health System Research Services, Tacoma, Washington
- Canada (7):
  - University of Calgary Foothills Medical Center, Calgary, Alberta
  - Vancouver Island Health Research Centre, Victoria, British Columbia
  - Health Sciences Centre, University of Manitoba, Winnepeg, Manitoba
  - Kingston General Hospital, Kingston, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - Centre de Sante et Services Sociaux de Chicoutimi, Chicoutimi, Quebec
  - Centre Hospitalier Regional de Trois-Rivieres, Trois-Rivières, Quebec

REFERENCES:
- [Derived] Montgomery DL, Matthews RP, Yee KL, Tobias LM, Dorr MB, Wrishko RE. Assessment of Bezlotoxumab Immunogenicity. Clin Pharmacol Drug Dev. 2020 Apr;9(3):330-340. doi: 10.1002/cpdd.729. Epub 2019 Aug 14. PMID 31411386
- [Derived] Gupta SB, Mehta V, Dubberke ER, Zhao X, Dorr MB, Guris D, Molrine D, Leney M, Miller M, Dupin M, Mast TC. Antibodies to Toxin B Are Protective Against Clostridium difficile Infection Recurrence. Clin Infect Dis. 2016 Sep 15;63(6):730-734. doi: 10.1093/cid/ciw364. Epub 2016 Jun 30. PMID 27365387
- [Derived] Lowy I, Molrine DC, Leav BA, Blair BM, Baxter R, Gerding DN, Nichol G, Thomas WD Jr, Leney M, Sloan S, Hay CA, Ambrosino DM. Treatment with monoclonal antibodies against Clostridium difficile toxins. N Engl J Med. 2010 Jan 21;362(3):197-205. doi: 10.1056/NEJMoa0907635. PMID 20089970

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inpatients and outpatients diagnosed with laboratory confirmed C. difficile disease whose physicians had opted to treat with standard of care (SOC) antibiotics, metronidazole by mouth (po)/ Intravenous (IV) or vancomycin po. A patient is considered eligible to participate in the study if a stool sample collected within 14 days of enrollment was positive by either the hospital/reference microbiology laboratory test or the rapid diagnostic test.
Pre-assignment Details: Prior to enrollment, patients had to meet the study definition of disease which allowed the inclusion of patients with moderate to severe diarrhea or colitis with or without accompanying systemic symptoms/signs (such as fever, nausea, anorexia, leukocytosis, abdominal pain, cramping or discomfort) whose disease was likely to continue for at least a few days after study enrollment.
Period: Overall Study
Arm/Group | GS-CDA1/MDX-1388 | Placebo
Started | 101 | 99
Completed | 92 | 86
Not Completed | 9 | 13
Not completed — Death | 7 | 8
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: 200 subjects who met the eligibility criteria and signed the informed consent randomized to receive study treatment: 101 in the GS-CDA1 and MDX-1388 (Monoclonal antibody (Mab)) treatment group and 99 in the placebo treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | GS-CDA1/MDX-1388 | Placebo | Total
Number analyzed (Participants) | 101 | 99 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (16.24) | 64 (15.02) | 64 (15.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 71 | 132
  Male | 40 | 28 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 97 | 93 | 190
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 91 | 84 | 175
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 9 | 13
A modified Horn's index for severity of underlying disease [Median (Full Range); unit: Scores on a severity scale] — The severity of underlying illness of the patient at the time of screening assessed by investigator or study nurse using a modified Horn's index. Horn's index graded on a scale of 1-3 from least to most severe. A patient with a score of 4 (catastrophic, life-threatening illness) at the time of screening is ineligible
  Scores on a severity scale | 2 [1 to 4] | 2 [1 to 4] | 2 [1 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrence of Clostridium Difficile Associated Disease (CDAD)
Description: Determine if the addition of C. difficile toxin A and toxin B human monoclonal anti-toxin antibodies to standard of care treatment reduces the number of subjects with recurrent CDAD compared to standard of care and placebo. Standard of care treatment is defined as receipt of either metronidazole by mouth or parenterally or receipt of vancomycin by mouth with a standard duration of treatment defined as 10 - 14 days (+ 2 days)). Recurrence of CDAD is defined as the development of a new episode of C. difficile disease associated with a positive C. difficile stool toxin(s) test after the resolution of prior episode and after discontinuation of SOC treatment.
Time Frame: Day 0 to Day 84
Population: 200 subjects who met the eligibility criteria and signed the informed consent and received standard of care treatment randomized 1:1 treatment allocation to receive study treatment: 101 subjects in the GS-CDA1/MDX-1388 (Monoclonal antibody (Mab)) treatment group and 99 subjects in the placebo treatment group
Measure: Count of Participants; unit: Participants
Arm/Group | GS-CDA1/MDX-1388 | Placebo
Number analyzed (Participants) | 101 | 99
Participants | 7 | 25

2. Secondary Outcome: Safety and Tolerability of Study Treatment by the Number of Adverse Events Reported
Description: Safety and tolerability of a C. difficile toxin A human monoclonal antibody combined with a human monoclonal antibody to C. difficile toxin B in patients receiving standard of care treatment for C. difficile associated disease (CDAD) compared to those patients receiving standard of care and placebo reporting system organ class (SOC) MedDRA V.9.0
Time Frame: Day 0 to Day 84
Population: as for outcome 1
Measure: Number; unit: Adverse Events
Arm/Group | GS-CDA1/MDX-1388 | Placebo
Number analyzed (Participants) | 101 | 99
Adverse Events
  Blood And Lymphatic System Disorders | 30 | 41
  Cardiac Disorders | 13 | 20
  Ear and Labyrinth | 3 | 3
  Endocrine Disorders | 0 | 1
  Eye Disorder | 7 | 7
  Gastrointestinal Disorders | 312 | 395
  General Disorders | 91 | 128
  Hepatobiliary Disorders | 1 | 1
  Immune Disorders | 1 | 0
  Infections And Infestations | 68 | 83
  Injury, Poisoning And Procedural Complications | 9 | 19
  Investigations | 18 | 30
  Metabolism And Nutrition Disorders | 55 | 128
  Musculoskeletal And Connective Tissue Disorders | 37 | 46
  Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps) | 3 | 1
  Nervous System Disorders | 61 | 79
  Psychiatric Disorders | 11 | 36
  Renal And Urinary Disorders | 9 | 9
  Reproductive System And Breast Disorders | 6 | 1
  Respiratory, Thoracic And Mediastinal Disorders | 36 | 61
  Skin And Subcutaneous Tissue Disorders | 27 | 17
  Surgical And Medical Procedures | 4 | 3
  Vascular Disorders | 9 | 19

3. Secondary Outcome: Time to Resolution of Initial CDAD Episode
Description: Determine if the addition of a C. difficile toxin A human monoclonal antibody combined with C. difficile toxin B human monoclonal antibody to standard of care treatment reduces the time to resolution of diarrhea in patients with CDAD compared to those patients receiving standard of care and placebo. Resolution of CDAD is defined as the cessation of diarrhea for at least two consecutive days.
Time Frame: Day 0 to Day 84
Population: 200 subjects who met the eligibility criteria and signed the informed consent and received standard of care treatment were randomized 1:1 treatment allocation to receive study treatment: 101 subjects in the GS-CDA1/MDX-1388 (Monoclonal antibody (Mab)) treatment group and 99 subjects in the placebo treatment group
Measure: Median (Full Range); unit: Days
Arm/Group | GS-CDA1/MDX-1388 | Placebo
Number analyzed (Participants) | 101 | 99
Days | 3 [0 to 84] | 3 [0 to 58]

4. Secondary Outcome: Number of Patients With Standard of Care Treatment Failure
Description: Determine if the addition of a C. difficile toxin A human monoclonal antibody combined with C. difficile toxin B human monoclonal antibody to standard of care treatment reduces the number of patients who experience standard of care treatment failure compared to those patients receiving standard of care and placebo. Standard of care treatment failure is defined as (i) recurrence of diarrhea (after it had initially resolved) while on SOC treatment during the first 14 days, or (ii) change in SOC treatment (i.e., antibiotics given), or (iii) diarrhea episode lasting ≥14 days while on SOC treatment.
Time Frame: Day 0 to Day 84
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | GS-CDA1/MDX-1388 | Placebo
Number analyzed (Participants) | 101 | 99
Participants | 21 | 24

5. Secondary Outcome: Number of Patients With Severe Initial C. Difficile Disease
Description: Determine if the addition of a C. difficile toxin A human monoclonal antibody combined with C. difficile toxin B human monoclonal antibody to standard of care treatment reduces the number of patients with severe C. difficile disease compared to those patients receiving standard of care and placebo. Severe initial disease is defined as ≥ 5 unformed stools/day for 2 consecutive days from day 1 to the end of the initial episode of diarrhea and discontinuation of SOC.
Time Frame: Day 0 to Day 84
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | GS-CDA1/MDX-1388 | Placebo
Number analyzed (Participants) | 101 | 99
Participants | 29 | 37

6. Secondary Outcome: Antibody Concentrations to Toxin A and to Toxin B Between Treatment Groups
Description: Antibody concentrations to Toxin A and to Toxin B in those patients receiving C. difficile toxin A human monoclonal antibody combined with C. difficile toxin B human monoclonal antibody and standard of care treatment to those patients receiving standard of care and placebo
Time Frame: Day 0 to Day 84
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: AUC0-∞ (hours x μg/ml)
Arm/Group | GS-CDA1/MDX-1388 | Placebo
Number analyzed (Participants) | 101 | 99
AUC0-∞ (hours x μg/ml)
  GS-CDA1 (Toxin A) | 115197.1 (37546.90) | NA (NA) — The majority of subjects in the placebo group had low or no detectable endogenous antibodies against either toxin.
  MDX-1388 (Toxin B) | 98540.9 (129413.74) | NA (NA) — The majority of subjects in the placebo group had low or no detectable endogenous antibodies against either toxin.

ADVERSE EVENTS:
Time Frame: Adverse events assessed from Day 0 through Day 84
Description: Adverse events assessed by interim medical history reviews, targeted physical assessments and clinical laboratory testing. Abnormal laboratory values constituted adverse events only if they induced clinical signs or symptoms or required new treatment or change in current therapy. Solicited adverse events included the occurrence of fever, chills, rash, joint pain or swelling, shortness of breath, headache, fatigue, or hives during the infusion and/or in the post-infusion period
Arm/Group | GS-CDA1/MDX-1388 | Placebo
All-Cause Mortality (participants affected / at risk) | 7/101 | 8/99
Serious Adverse Events (participants affected / at risk) | 18/101 | 28/99
Other Adverse Events (participants affected / at risk) | 100/101 | 99/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GS-CDA1/MDX-1388 (N=101) | Placebo (N=99)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 3 (3)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 2 (2)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 2 (3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 2 (2)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 5 (6)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 2 (2)
ASTHENIA (General disorders) | 1 (1) | 1 (1) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
CHEST PAIN (General disorders) | 0 (0) | 1 (1) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
LOWER EXTREMITY MASS (General disorders) | 1 (1) | 0 (0) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (1) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
PYREXIA (General disorders) | 0 (0) | 2 (2) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
SUDDEN DEATH (General disorders) | 1 (1) | 0 (0) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
HEPATITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 5 (5) | 7 (7)
INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LOBAR PNEUMONIA (Infections and infestations) | 1 (1) | 2 (2)
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 3 (3)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 4 (4)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
UROSEPSIS (Infections and infestations) | 1 (1) | 1 (1)
DIALYSIS DEVICE COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BLOOD CULTURE POSITIVE (Investigations) | 0 (0) | 1 (1)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
METABOLIC DISORDER (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 0 (0) | 1 (3)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (3)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COLECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
ILEOSTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 0 (0)
EMBOLISM (Vascular disorders) | 1 (1) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 7 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GS-CDA1/MDX-1388 (N=101) | Placebo (N=99)
ANAEMIA (Blood and lymphatic system disorders) | 4 (5) | 5 (5)
COAGULOPATHY (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 15 (21) | 18 (27)
NEUTROPHILIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
SPLENOMEGALY (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 1 (2)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 1 (2)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1) | 2 (2)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDIAL HAEMORRHAGE (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDITIS (Cardiac disorders) | 1 (1) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 2 (2)
EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 0 (0)
EXTERNAL EAR INFLAMMATION (Ear and labyrinth disorders) | 0 (0) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 1 (1) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
CONJUNCTIVITIS (Eye disorders) | 0 (0) | 1 (2)
CONJUNCTIVITIS ALLERGIC (Eye disorders) | 1 (1) | 0 (0)
DRY EYE (Eye disorders) | 1 (1) | 1 (2)
ECTROPION (Eye disorders) | 1 (1) | 0 (0)
EYE INFLAMMATION (Eye disorders) | 0 (0) | 1 (1)
KERATITIS (Eye disorders) | 1 (1) | 0 (0)
LACRIMATION INCREASED (Eye disorders) | 1 (1) | 0 (0)
OCULAR HYPERAEMIA (Eye disorders) | 1 (1) | 1 (1)
VISION BLURRED (Eye disorders) | 1 (1) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 2 (2) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 5 (5) | 6 (9)
ABDOMINAL PAIN (Gastrointestinal disorders) | 51 (109) | 45 (122)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ANAL FISSURE (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (2)
COELIAC DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 40 (69) | 55 (104)
DIVERTICULUM (Gastrointestinal disorders) | 0 (0) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 4 (6) | 3 (3)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ERUCTATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 3 (6) | 6 (10)
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 2 (2)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMATOCHEZIA (Gastrointestinal disorders) | 13 (17) | 10 (13)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 4 (5)
MUCOUS STOOLS (Gastrointestinal disorders) | 0 (0) | 1 (3)
NAUSEA (Gastrointestinal disorders) | 37 (65) | 42 (74)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 2 (2) | 1 (1)
PERIANAL ERYTHEMA (Gastrointestinal disorders) | 1 (1) | 1 (1)
PROCTALGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL FISSURE (Gastrointestinal disorders) | 1 (1) | 0 (0)
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
SWOLLEN TONGUE (Gastrointestinal disorders) | 0 (0) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 14 (18) | 11 (18)
ADVERSE DRUG REACTION (General disorders) | 1 (1) | 0 (0) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
ASTHENIA (General disorders) | 3 (4) | 8 (10) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
CHEST DISCOMFORT (General disorders) | 0 (0) | 4 (4) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
CHEST PAIN (General disorders) | 2 (2) | 3 (5) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
CHILLS (General disorders) | 2 (2) | 6 (7) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
DISCOMFORT (General disorders) | 1 (4) | 0 (0) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
FATIGUE (General disorders) | 26 (47) | 22 (50) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
GENERALISED OEDEMA (General disorders) | 0 (0) | 1 (1) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
HERNIA PAIN (General disorders) | 0 (0) | 1 (1) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
IMPLANT SITE EFFUSION (General disorders) | 1 (1) | 0 (0) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
INFLAMMATION (General disorders) | 1 (1) | 0 (0) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
INFUSION SITE SWELLING (General disorders) | 0 (0) | 1 (1) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
OEDEMA (General disorders) | 2 (3) | 1 (1) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
OEDEMA PERIPHERAL (General disorders) | 6 (6) | 5 (6) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
PAIN (General disorders) | 2 (2) | 7 (7) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
PITTING OEDEMA (General disorders) | 1 (1) | 0 (0) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
PYREXIA (General disorders) | 9 (14) | 18 (30) — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
LIVER DISORDER (Hepatobiliary disorders) | 0 (0) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ARTHRITIS INFECTIVE (Infections and infestations) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
BRONCHIECTASIS (Infections and infestations) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
CANDIDIASIS (Infections and infestations) | 2 (2) | 1 (1)
CELLULITIS (Infections and infestations) | 2 (2) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2 (3) | 9 (10)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1)
CYSTITIS BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
EYE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
FUNGAL INFECTION (Infections and infestations) | 2 (5) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
HERPES SIMPLEX (Infections and infestations) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1)
IMPETIGO (Infections and infestations) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 2 (2) | 0 (0)
LABYRINTHITIS (Infections and infestations) | 1 (1) | 0 (0)
LARYNGITIS (Infections and infestations) | 1 (1) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 1 (1) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 6 (6) | 1 (1)
ORAL CANDIDIASIS (Infections and infestations) | 2 (2) | 2 (2)
PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (3) | 5 (5)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1)
RHINITIS (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 2 (3) | 1 (3)
TINEA INFECTION (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (5) | 5 (5)
URINARY TRACT INFECTION (Infections and infestations) | 8 (9) | 16 (18)
URINARY TRACT INFECTION FUNGAL (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (1)
VAGINAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1)
VAGINAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 1 (1) | 1 (2)
ARTERIOVENOUS FISTULA SITE HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ARTERIOVENOUS FISTULA THROMBOSIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BACK INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
EXCORIATION (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 4 (5)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TOOTH INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE ABNORMAL (Investigations) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 1 (1)
ANTIMICROBIAL SUSCEPTIBILITY TEST RESISTANT (Investigations) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE ABNORMAL (Investigations) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 2 (2)
BACTERIAL CULTURE (Investigations) | 1 (1) | 0 (0)
BACTERIAL CULTURE POSITIVE (Investigations) | 0 (0) | 1 (1)
BLOOD ALBUMIN DECREASED (Investigations) | 1 (1) | 1 (1)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD MAGNESIUM DECREASED (Investigations) | 1 (1) | 2 (2)
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 (0) | 1 (1)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 1 (2)
BLOOD UREA DECREASED (Investigations) | 0 (0) | 1 (1)
BLOOD UREA INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD URINE PRESENT (Investigations) | 2 (2) | 0 (0)
BODY TEMPERATURE INCREASED (Investigations) | 1 (1) | 0 (0)
CARDIAC MURMUR (Investigations) | 1 (1) | 1 (1)
CULTURE URINE POSITIVE (Investigations) | 0 (0) | 1 (1)
ELECTROCARDIOGRAM ST SEGMENT ABNORMAL (Investigations) | 0 (0) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 1 (1)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 2 (2) | 2 (2)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 2 (2)
OCCULT BLOOD (Investigations) | 0 (0) | 1 (1)
PLATELET COUNT INCREASED (Investigations) | 0 (0) | 1 (1)
PROTHROMBIN TIME PROLONGED (Investigations) | 0 (0) | 1 (1)
URINE ANALYSIS ABNORMAL (Investigations) | 1 (1) | 0 (0)
URINE OUTPUT DECREASED (Investigations) | 0 (0) | 1 (1)
VITAMIN D DECREASED (Investigations) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 2 (2)
ANOREXIA (Metabolism and nutrition disorders) | 20 (28) | 42 (55)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 7 (8)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
GOUT (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
HYPOCHLORAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 9 (9) | 13 (18)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 5 (6)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MALNUTRITION (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (9) | 10 (13)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (10)
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 6 (10) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SACRAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
LIPOSARCOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PYOGENIC GRANULOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BALANCE DISORDER (Nervous system disorders) | 1 (1) | 1 (1)
BURNING SENSATION (Nervous system disorders) | 2 (2) | 0 (0)
DIZZINESS (Nervous system disorders) | 12 (13) | 16 (19)
DYSGEUSIA (Nervous system disorders) | 1 (1) | 3 (3)
HEADACHE (Nervous system disorders) | 23 (35) | 29 (38)
LETHARGY (Nervous system disorders) | 0 (0) | 2 (2)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 1 (1)
MIGRAINE (Nervous system disorders) | 1 (5) | 2 (5)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 0 (0)
PARKINSON'S DISEASE (Nervous system disorders) | 0 (0) | 1 (1)
SINUS HEADACHE (Nervous system disorders) | 1 (1) | 1 (3)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1)
TREMOR (Nervous system disorders) | 1 (1) | 1 (1)
AGITATION (Psychiatric disorders) | 1 (1) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1) | 8 (13)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 1 (1)
DELIRIUM (Psychiatric disorders) | 1 (1) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 5 (5)
HALLUCINATION (Psychiatric disorders) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 3 (5) | 10 (12)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 1 (1)
NIGHTMARE (Psychiatric disorders) | 1 (1) | 0 (0)
NOCTIPHOBIA (Psychiatric disorders) | 1 (1) | 0 (0)
OBSESSIVE-COMPULSIVE DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
BLADDER PAIN (Renal and urinary disorders) | 1 (1) | 1 (1)
BLADDER SPASM (Renal and urinary disorders) | 0 (0) | 1 (1)
DYSURIA (Renal and urinary disorders) | 0 (0) | 2 (2)
NEPHROGENIC DIABETES INSIPIDUS (Renal and urinary disorders) | 1 (1) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1)
POLLAKIURIA (Renal and urinary disorders) | 2 (2) | 0 (0)
POLYURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
PYURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL DISORDER (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 1 (1)
URINARY BLADDER POLYP (Renal and urinary disorders) | 1 (1) | 0 (0)
BREAST PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0)
DYSMENORRHOEA (Reproductive system and breast disorders) | 2 (3) | 0 (0)
FIBROCYSTIC BREAST DISEASE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
GENITAL PRURITUS FEMALE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
GYNAECOMASTIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (13)
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (6)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPERVENTILATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOCAPNIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
OROPHARYNGEAL SWELLING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (5)
PICKWICKIAN SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
UPPER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
COLD SWEAT (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HYPOTRICHOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 8 (11) | 3 (3)
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
CHOLECYSTECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
EYE OPERATION (Surgical and medical procedures) | 0 (0) | 1 (1)
HAEMORRHOID OPERATION (Surgical and medical procedures) | 1 (1) | 0 (0)
OPEN REDUCTION OF FRACTURE (Surgical and medical procedures) | 1 (1) | 0 (0)
PARENTERAL NUTRITION (Surgical and medical procedures) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
FLUSHING (Vascular disorders) | 1 (1) | 0 (0)
HOT FLUSH (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 2 (2) | 5 (6)
HYPOTENSION (Vascular disorders) | 1 (1) | 4 (4)
STEAL SYNDROME (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less